CLINICAL TRIAL: NCT05663268
Title: Efficacy and Safety of Infliximab Biosimilar in the Treatment of Resistant Hidradenitis Suppurativa
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Hira Tariq, Principal Investigator, Services Institute of Medical Sciences, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2022/101/SIMS
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; Infliximab biosimilar; Efficacy; safety
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — CT-P13

STUDY DESIGN:
Intervention Model Description: Adult patients of either gender suffering from Hidradenitis suppurativa resistant to conventional therapies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients of Hidradenitis suppurativa resistant to conventional therapy (Experimental): injection Infliximab-dyyb biosimilar (according to weight, single injection of 120mg if weight <80kg, 2 injections if weight > 80kg) will be injected subcutaneously at week 0,1, 2,3,4, and then fortnightly till 24 weeks.
  Interventions: Biological: Infliximab-dyyb biosimilar

INTERVENTIONS:
Biological: Infliximab-dyyb biosimilar — Remsima for subcutaneous injection is a biosimilar monoclonal antibody of infliximab-dyyb that inhibits the activity of tumour necrosis factor (TNF)-alpha.
  Other Names: Remsima (infliximab-dyyb biosimilar)

SUMMARY:
The aim of this clinical trial is to assess the efficacy and safety of Infliximab-dyyb biosimilar in patients of resistant Hidradenitis suppurativa. The main question it aims to answer are:

* how effective is infliximab biosimilar in treating resistant Hidradentis suppurativa
* Is infliximab biosimilar safe in these patients Patients will receive weekly injections of Infliximab Biosimilar Remsima, according to weight, for first 4 weeks, and then fortnightly for next 24 weeks. Patients will be followed up at 4, 14 and 24 weeks for assessment of safety and efficacy

DETAILED DESCRIPTION:
The aim of this clinical trial is to assess the efficacy and safety of Infliximab-dyyb biosimilar in patients of resistant Hidradenitis suppurativa. The main question it aims to answer are:

* how effective is infliximab biosimilar in treating resistant Hidradentis suppurativa
* Is infliximab biosimilar safe in these patients Patients will receive weekly injections of Infliximab Biosimilar Remsima, according to weight, for first 4 weeks, and then fortnightly for next 24 weeks. Patients will be followed up at 4, 14 and 24 weeks for assessment of safety and efficacy.

Pre and post treatment HiSCR, IHS4, DLQI scores and photos will be taken for comparison at week 0, 4, 14 and 24. Details will be entered on predesigned proforma DATA ANALYSIS PROCEDURE: Data will be entered and analyzed using SPSS 20. Data will be stratified for role of effect modifiers.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Hidradenitis suppurativa resistant to conventional therapy

Exclusion Criteria:

* Immunocompromised patients
* Patients with connective tissue disorders
* patients having chronic infections like heapatitis, HIV or Tuberculosis
* Pregnant or lactating mothers
* hypersensitivity to biologics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response (HiSCR) | 24 weeks
  50% reduction in score
Dermatology Life Quality Index (DLQI) | 24 weeks
  50% reduction

CONTACTS AND LOCATIONS:
Overall Officials: Hira Tariq, FCPS Derma, Principal Investigator — Services Institute of Medical Sciences, Pakistan
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fernandez-Vozmediano JM, Armario-Hita JC. Infliximab for the treatment of hidradenitis suppurativa. Dermatology. 2007;215(1):41-4. doi: 10.1159/000102032. PMID 17587838
- [Result] Sullivan TP, Welsh E, Kerdel FA, Burdick AE, Kirsner RS. Infliximab for hidradenitis suppurativa. Br J Dermatol. 2003 Nov;149(5):1046-9. doi: 10.1111/j.1365-2133.2003.05663.x. PMID 14632813